CLINICAL TRIAL: NCT01472835
Title: Randomized, Cross-over Study Evaluating the Effect of Sedation on Pain Relief After Diagnostic Injections
Brief Title: Effect of Sedation on Diagnostic Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven P. Cohen, Professor, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00045905
Record Dates: First submitted 2011-04-25; First posted 2011-11-17 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-10

CONDITIONS: Sacroiliac Joint Pain; Sympathetically Maintained Pain
Keywords: sedation; sensitivity; specificity; validity; diagnostic injection
MeSH Terms: conditions — Hypersensitivity | interventions — Midazolam; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sedation (Experimental): Pt will receive sedation with their procedure
  Interventions: Drug: Midazolam; Drug: Fentanyl
- Control (No Intervention): Patient will not receive sedation during procedure

INTERVENTIONS:
Drug: Midazolam — Used for anxiolysis
  Arms: Sedation
Drug: Fentanyl — Used for analgesia and as a sedative
  Arms: Sedation

SUMMARY:
Interventional pain procedures have diagnostic, prognostic and therapeutic value. It is well-documented that the reference standard for identifying a pain generator is a low-volume block performed with local anesthetic, with or without steroid. Many factors may increase the false positive (FP) rate of diagnostic and prognostic nerve blocks; however, the use of sedation is the most controversial and remediable. Proponents of sedation argue that it has little effect on the rate of positive diagnostic blocks, and may even reduce the false-negative rate. The purpose of this study is to determine the effect of intravenous sedation on pain relief and the "false-positive rate" after diagnostic nerve blocks.

DETAILED DESCRIPTION:
Sixty-eight patients with sacroiliac (SI) joint or sympathetically-maintained pain will be randomized in a crossover fashion to receive diagnostic nerve blocks either with or without intravenous sedation. Among those who obtain some benefit and return for a 2nd block, this 2nd procedure will be done with sedation if the first was done without sedation, and vice versa. Midazolam and fentanyl will be used for intravenous sedation, titrated to anxiolysis and analgesia. Pain scores (0-10 numerical rating scale, or NRS) and an activity log will be recorded over the 8-hours following the blocks via a pain diary. The first follow-up visit will be 4 weeks after the procedure. Patients who obtain some benefit but continue to report significant pain or who might otherwise benefit from a repeat procedure will have this second procedure performed with sedation if no sedation was given for the first procedure, and without sedation if sedation was administered for the first procedure. The post-procedure pain data will be recorded in the same fashion as the initial nerve block. The second follow-up visit will be 4 weeks after the 2nd block.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain > 4 weeks but < 10 years in duration
* Suspected SI joint or sympathetically-maintained pain based on history and physical exam
* May benefit from a sacroiliac joint or sympathetic block
* Pain on 0-10 NRS scale > 3/10 in intensity

Exclusion Criteria:

* No previous interventional pain-alleviating injections for the same condition within the past 3 years
* Uncontrolled coagulopathy
* Pregnancy, which will be ruled out by a urine pregnancy test in women of childbearing age
* Allergy to contrast dye or amide local anesthetics
* Unstable medical or psychiatric condition (e.g. unstable angina, congestive heart failure or severe depression) that could preclude an optimal treatment response
* Systemic infection
* Age < 18 or > 75 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Cohen, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Blaustein Pain Treatment Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Cohen SP, Hurley RW. The ability of diagnostic spinal injections to predict surgical outcomes. Anesth Analg. 2007 Dec;105(6):1756-75, table of contents. doi: 10.1213/01.ane.0000287637.30163.a2. PMID 18042881
- [Derived] Cohen SP, Hameed H, Kurihara C, Pasquina PF, Patel AM, Babade M, Griffith SR, Erdek ME, Jamison DE, Hurley RW. The effect of sedation on the accuracy and treatment outcomes for diagnostic injections: a randomized, controlled, crossover study. Pain Med. 2014 Apr;15(4):588-602. doi: 10.1111/pme.12389. Epub 2014 Feb 13. PMID 24524866

RESULTS

PARTICIPANT FLOW:
Groups:
- Sedation: Pt will receive sedation with their 1st procedure, then a control procedure will be done without sedation
  sacroiliac joint injection: Patient will receive an injection into the sacroiliac joint with bupivacaine and corticosteroid with and without sedation. Since this is a crossover trial, patients will receive both "treatments".
  Sympathetic block: Sympathetic block with bupivacaine
  bupivacaine
  corticosteroid
- Control: Patient will not receive sedation during their 1st procedure, but receive sedation during the 2nd procedure
Period: Overall Study
Arm/Group | Sedation | Control
Started | 37 | 36
Completed | 35 | 36
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sedation: Pt will receive sedation with their 1st procedure and no sedation with their 2nd procedure
  sacroiliac joint injection: Patient will receive an injection into the sacroiliac joint with bupivacaine and corticosteroid with and without sedation. Since this is a crossover trial, patients will receive both "treatments".
  Sympathetic block: Sympathetic block with bupivacaine
  bupivacaine
  corticosteroid
- Control: Patient will not receive no sedation during their 1st procedure and sedation during their 2nd procedure
- Total: Total of all reporting groups
Arm/Group | Sedation | Control | Total
Number analyzed (Participants) | 37 | 36 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (16.1) | 50.3 (13.8) | 50.0 (15.0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 35 | 67
  >=65 years | 5 | 1 | 6
Gender [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 17 | 14 | 31
Region of Enrollment [Number; unit: participants]
  United States | 37 | 36 | 73

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: pain diary using 0-10 scale, with 0 being no pain and 10 being the worst pain imaginable
Time Frame: through 6 hours after injection
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control: Patient will not receive sedation during their 1st procedure but receive sedation during their 2nd procedure
Arm/Group | Sedation | Control
Number analyzed (Participants) | 36 | 36
units on a scale | 2.2 (2.3) | 3.4 (2.8)

2. Secondary Outcome: Pain Score
Description: 0-10 numerical rating scale (NRS) pain scale. 0 being no pain and 10 being the worst possible pain.
Time Frame: 1-month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sedation: Pt will receive sedation with their procedure
  sacroiliac joint injection: Patient will receive an injection into the sacroiliac joint with bupivacaine and corticosteroid with and without sedation. Since this is a crossover trial, patients will receive both "treatments".
  Sympathetic block: Sympathetic block with bupivacaine
  bupivacaine
  corticosteroid
Arm/Group | Sedation | Control
Number analyzed (Participants) | 36 | 36
units on a scale | 5.1 (2.9) | 5.6 (2.8)

3. Secondary Outcome: Procedure-related Pain Score
Description: 0-10 pain scale, with 0 being no pain and 10 being the worst pain imaginable
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control: Patient will not receive sedation during the 1st procedure, but receive sedation during their 2nd procedure
Arm/Group | Sedation | Control
Number analyzed (Participants) | 36 | 36
units on a scale | 3.1 (2.8) | 5.5 (2.7)

4. Secondary Outcome: Oswestry Disability Index
Description: Measure of functional capacity on a scale ranging from 0% to 100%, with 0% signifying no disability
Time Frame: 1-month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sedation | Control
Number analyzed (Participants) | 36 | 36
units on a scale | 34.8 (14.6) | 40.6 (17.9)

5. Secondary Outcome: Satisfaction
Description: 5-point Likert scale. The scale is from 1-5. 1 being very unsatisfied and 5 being very satisfied.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sedation | Control
Number analyzed (Participants) | 36 | 36
units on a scale | 4.0 (1.1) | 3.6 (1.4)

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Sedation: Pt received sedation with their procedure
  sacroiliac joint injection: Patient will receive an injection into the sacroiliac joint with bupivacaine and corticosteroid with and without sedation. Since this is a crossover trial, patients will receive both "treatments".
  Sympathetic block: Sympathetic block with bupivacaine
  bupivacaine
  corticosteroid
- Control: Patient did not receive sedation during procedure
Arm/Group | Sedation | Control
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/36
Other Adverse Events (participants affected / at risk) | 3/37 | 6/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sedation (N=37) | Control (N=36)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) — Less than 1 day
dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Less than 1 day
Headache (Nervous system disorders) | 1 (1) | 1 (1) — Less than 1 day
Worse pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Less than 1 week
Weakness (Nervous system disorders) | 0 (0) | 1 (1) — Less than 1 day
Dizziness (General disorders) | 0 (0) | 1 (1) — Less than 1 day

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No